CLINICAL TRIAL: NCT06104449
Title: A Phase 1 Clinical Study to Investigate the Safety and Pharmacokinetics of MK-5684 in Japanese Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: A Study of Opevesostat (MK-568)4 in Japanese Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC) (MK-5684-005)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5684-005; MK-5684-005 (Other: MSD); jRCT2031230431 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Prostatic Neoplasms; Metastatic Castration-Resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dexamethasone; Calcium Dobesilate; fludrocortisone acetate; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Opevesostat (Experimental): Participants receive opevesostat 5 mg by oral tablets twice daily plus dexamethasone 1.5 mg by oral tablets and fludrocortisone acetate 0.1 mg oral tablet once daily continuously until progression. Hydrocortisone up to 100 mg oral dose will also be provided to participants for use as rescue medication.
  Interventions: Drug: Opevesostat; Drug: Dexamethasone; Drug: Fludrocortisone acetate; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Opevesostat — Tablets to be taken orally.
  Other Names: MK-5684
Drug: Dexamethasone — Tablets to be taken orally.
  Other Names: Decadron
Drug: Fludrocortisone acetate — Tablet to be taken orally.
Drug: Hydrocortisone — Tablets to be taken orally as a recue medication.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of opevesostat in the treatment of Japanese men with metastatic castration-resistant prostate cancer (mCRPC) previously treated with Next Generation Hormonal Agent (NHA) and taxane-based chemotherapy.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has histologically- or cytologically-confirmed adenocarcinoma of the prostate without small cell histology
* Has current evidence of metastatic disease documented by either bone lesions on bone scan and/or soft tissue disease by computed tomography/magnetic resonance imaging (CT/MRI)
* Has ongoing androgen deprivation with serum testosterone <50 ng/dL (<1.7 nmol/L)
* Participants receiving bone anti-resorptive therapy (including, but not limited to bisphosphonate or denosumab) must have been on stable doses for ≥4 weeks prior to the start of study intervention.
* Has progressed on or after treatment with at least 1 line of NHAs in metastatic hormone-sensitive prostate cancer (mHSPC) or in castration-resistant prostate cancer (CRPC) for a minimum of 12 weeks (e.g. abiraterone, enzalutamide, darolutamide, apalutamide), and with at least 1 line of taxane-based chemotherapy in mHSPC or in CRPC, or ineligibility for chemotherapy
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 10 days prior to allocation
* If capable of producing sperm, participant must agree to the following during the study treatment period and for at least 7 days after the last dose of opevesostat: Refrain from donating sperm, plus EITHER be abstinent OR must agree to use male condom.

Exclusion Criteria:

* Has a history of pituitary dysfunction
* Has brain metastases
* History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 3 years
* Has an active or uncontrolled autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs)
* Has an active infection or other medical condition that would make corticosteroid contraindicated
* Has serious persistent infection within 2 weeks prior to the start of the study intervention
* Participants on an unstable dose of thyroid hormone therapy within 6 months prior to the start of the study intervention
* Has poorly controlled diabetes mellitus
* Hypotension: systolic blood pressure (BP) < 110 mmHg, or uncontrolled hypertension: systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg, in 2 out of 3 recordings with optimized antihypertensive therapy
* Has active or unstable cardio/cerebro-vascular disease, including thromboembolic event
* Is unable to swallow orally administered medication or known gastrointestinal (GI) disease or GI procedure that may interfere with absorption of study intervention
* Has undergone major surgery including local prostate intervention (excluding prostate biopsy) within 28 days prior to the start of the study intervention and not adequately recovered from the toxicities and/or complications
* Has received aldosterone antagonist (e.g. spironolactone, eplerenone) and phenytoin within 4 weeks prior to the start of the study intervention
* Has received radiotherapy within 4 weeks prior to the start of the study intervention, or radiation related toxicities, requiring corticosteroids
* Has received chemotherapy within the last 4 weeks (2 weeks for oral or weekly chemotherapy; 6 weeks for nitrosoureas and mitomycin C) prior to the start of the study intervention
* Has received prior enzalutamide and apalutamide within 3 weeks, or abiraterone and darolutamide within 2 weeks prior to the start of the study intervention
* Systemic use of the following medications within 2 weeks prior to the start of study intervention: strong cytochrome P450 (CYP)3A4 inducers: e.g., carbamazepine, rifampicin, phenobarbital, phenytoin, St John's Wort) and strong CYP3A4 inhibitors: e.g., itraconazole, ketoconazole, posaconazole, voriconazole, clarithromycin, telithromycin, grapefruit juice
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed.
* Has used herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (eg, saw palmetto) within 4 weeks prior to the start of the study intervention
* Has received treatment with 5-α reductase inhibitors (eg, finasteride or dutasteride), estrogens, and/or cyproterone within 4 weeks prior to the start of the study intervention
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* History of human immunodeficiency virus (HIV) infection
* Has a history of Hepatitis B or active Hepatitis C virus
* Has a "superscan" bone scan
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the start of the study intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Dose-limiting Toxicity (DLT) as Assessed Using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 by the Investigator | Up to 28 days
  The following events, if considered drug related by the Investigator, will be considered a DLT: Grade 4 hematologic toxicity lasting ≥7 days, except anemia and thrombocytopenia; Grade 3 nausea, vomiting, diarrhea or fatigue lasting >3 days despite optimal supportive care; other nonhematologic grade ≥3 toxicities of any duration (not laboratory); Grade ≥3 nonhematologic laboratory abnormality (if certain criteria are met); febrile neutropenia Grade 3 or Grade 4; missing >25% of opevesostat doses as a result of drug-related AE(s) during the first 28 days; Grade 5 toxicity. The number of participants who experience a DLT will be presented.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 24 months
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 24 months
  An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of opevesostat | Day 1, Day 8, Day 29, and at first visit after the last dose of opevesostat (up to approximately 24 months)
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the Cmax.
Time to Maximum Plasma Concentration (Tmax) of opevesostat | Day 1, Day 8, Day 29, and at first visit after the last dose of opevesostat (up to approximately 24 months)
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the Tmax.
Area Under the Curve from Time 0 to 12 hours postdose (AUC0-12) of opevesostat | Day 1, Day 8, Day 29, and at first visit after the last dose of opevesostat (up to approximately 24 months)
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the AUC0-12.
Apparent Volume of Distribution (Vz/F) of opevesostat | Day 1, Day 8, Day 29, and at first visit after the last dose of opevesostat (up to approximately 24 months)
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the Vz/F.
Oral Clearance (CL/F) of opevesostat | Day 1, Day 8, Day 29, and at first visit after the last dose of opevesostat (up to approximately 24 months)
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the CL/F.
Half-Life (t½) of opevesostat | Day 1, Day 8, Day 29, and at first visit after the last dose of opevesostat (up to approximately 24 months)
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine the t½.
Prostate-specific Antigen (PSA) response | Up to approximately 24 months
  Percentage of participants in the analysis population who have a reduction in PSA level of ≥50% measured twice ≥3 weeks apart.
Time to Prostate-specific Antigen (PSA) Progression | Up to approximately 24 months
  Time from first dose of study drug to PSA progression. PSA progression date is defined as the date of 1) ≥25% increase and ≥2 ng/mL above the nadir, confirmed by a second value ≥3 weeks later if there is PSA decline from baseline, or 2) ≥25% increase and ≥2 ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline.
Radiographic Progression-free Survival (rPFS) Per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator | Up to approximately 24 months
  Time from first dose of study drug to radiographic progression, or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) Per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator | Up to approximately 24 months
  Percentage of participants in the analysis population who have a best overall response of either confirmed Complete Response (CR) or a confirmed Partial Response (PR) per PCWG-modified RECIST 1.1.
Duration of Response (DOR) Per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator | Up to approximately 24 months
  Time from first documented evidence of confirmed Complete Response (CR) or Partial Response (PR) per PCWG-modified RECIST 1.1 until disease progression or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 24 months
  Time from first dose of study intervention to death due to any cause.
Blood Concentrations of Steroids | Day 1, Day 8, Day 29, Day 85, and at first visit after the last dose of opevesostat (up to approximately 24 months)
  Blood samples collected at multiple timepoints after the administration of opevesostat will be used to determine the blood concentrations of steroids.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- Japan (3):
  - National Cancer Center Hospital East ( Site 0001), Kashiwa, Chiba
  - Toho University Sakura Medical Center ( Site 0003), Sakura, Chiba
  - Yokohama City University Medical Center ( Site 0002), Yokohama, Kanagawa

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com